CLINICAL TRIAL: NCT07373392
Title: Effects of LP-LDL® on Lipid Metabolism, Glycemic Control, Inflammatory Markers, and Cognitive Function in Individuals With Prediabetes and Diabetes Mellitus (Type 1 and Type 2)
Brief Title: Effects of LP-LDL® on Lipid Metabolism, Glycemic Control, Inflammatory Markers, and Cognitive Function in Individuals With Prediabetes and Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Steno Diabetes Center Nordjylland (Other); ProBiotix Health Plc. (Unknown)
Responsible Party: Principal Investigator, Hiva Alipour, Associate Professor, Department of Health Science and Technology, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-20250029
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabete Type 1; Diabete Type 2; Prediabetes
Keywords: Prediabetes; Type 1 Diabetes; Type 2 Diabetes; Dyslipidemia; Hypercholesterolemia; Metabolic dysfunction; Insulin resistance; Probiotics; LP-LDL; Lactobacillus plantarum; Lactobacillus plantarum ECGC 13110402; Dietary supplement; Microbiome modulation; LDL cholesterol; Cardiometabolic health
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus, Type 1; Dyslipidemias; Hypercholesterolemia; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LP-LDL® (Active Treatment) (Active Comparator): Product: LP-LDL® (Lactobacillus plantarum ECGC 13110402) Dose: ≥4×10⁹ CFU, one capsule daily Duration: 12 weeks
  Interventions: Dietary Supplement: Lactobacillus plantarum ECGC 13110402
- Placebo (Placebo Comparator): An identical capsule without an active bacterial strain Dose: one capsule daily Duration: 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum ECGC 13110402 — LP-LDL® (Lactobacillus plantarum ECGC 13110402) is a probiotic dietary supplement provided in a capsule containing a minimum of 4 × 10⁹ CFU of the viable bacterial strain at the time of release. Each active capsule contains 50 mg of freeze-dried Lactobacillus plantarum ECGC 13110402, blended with 165 mg of corn starch and 25 mg of microcrystalline cellulose as excipients. Participants assigned to the active arm will take one capsule orally once daily for 12 weeks.
  Other Names: LP-LDL
  Arms: LP-LDL® (Active Treatment)
Dietary Supplement: Placebo — The placebo consists of an identical capsule containing only the excipients (215 mg corn starch and 25 mg microcrystalline cellulose) without any live bacteria. Active and placebo capsules are identical in appearance, packaging, labeling, and handling to maintain blinding. All products are manufactured, blended, encapsulated, blind-labeled, and packaged under GMP conditions by ProBiotix Health.
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial investigates the effects of the probiotic LP-LDL® (Lactobacillus plantarum ECGC 13110402) on lipid metabolism, glycemic control, inflammatory biomarkers, and cognitive function in adults with prediabetes, type 1 diabetes, or type 2 diabetes who also exhibit elevated cholesterol or triglyceride levels.

A total of 210 participants will be enrolled across three parallel sub-studies:

* Type 1 diabetes (n = 76)
* Type 2 diabetes (n = 54)
* Prediabetes (n = 80)

Participants will be randomized 1:1 to receive LP-LDL® or matching placebo once daily for 12 weeks, followed by a 4-week washout period. Study assessments include fasting blood tests (lipids, glucose, HbA1c, liver enzymes, inflammatory markers), cognitive testing (ACE-III), blood pressure, anthropometry, and stool measurements (microbiome, bile acids, fecal fat).

Exploratory analyses include bile acid metabolism, microbiome profiling (16S rRNA), and gene expression of cholesterol transporters ABCG5/ABCG8.

The study aims to determine whether LP-LDL® can improve cardiometabolic profiles and cognitive outcomes in these populations, and to clarify the mechanistic pathways underlying metabolic dysfunction, inflammation, and gut-brain communication.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Prediabetes (FPG 100-125 mg/dL or HbA1c 42-47 mmol/mol), or Type 1 or Type 2 diabetes
* Elevated cholesterol or triglycerides (TC ≥200 mg/dL, LDL 130-189 mg/dL, or TG >150 mg/dL)
* Either no lipid-lowering medication or stable dose for ≥4 weeks
* Able to swallow capsules and understand Danish
* Willing to maintain lifestyle habits and provide stool and blood samples

Exclusion Criteria:

* Antibiotic use in the past 3 months
* Severe dyslipidemia (>500 mg/dL triglycerides)
* Significant liver, kidney, thyroid disease
* Pregnancy or breastfeeding
* GI surgery or chronic GI disease (IBD, IBS, Crohn's disease)
* Long-term medications influencing lipid/glucose metabolism (except approved antidiabetic medications)
* Participation in another trial within 3 months
* Capsule intake <80%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in lipid profile (total cholesterol, LDL, HDL, triglycerides) | Baseline, Week 6, Week 12, Week 16

SECONDARY OUTCOMES:
Fasting blood glucose | Baseline, Week 6, Week 12, Week 16
HbA1c | Baseline, Week 6, Week 12, Week 16
Apolipoprotein A-I and B levels | Baseline, Week 6, Week 12, Week 16
Blood pressure | Baseline, Week 6, Week 12, Week 16
Liver enzymes (ALT, AST, ALP) | Baseline, Week 6, Week 12, Week 16
Cognitive function (Addenbrooke's Cognitive Examination-III (ACE-III)) | Baseline, Week 6, Week 12, Week 16
CRP | Baseline, Week 6, Week 12, Week 16
IL-6 | Baseline, Week 6, Week 12, Week 16

OTHER OUTCOMES:
Bile acid metabolites (LC-MS/GC-MS) | Baseline, Week 6, Week 12, Week 16
Fecal microbiome composition (16S rRNA) | Baseline, Week 6, Week 12, Week 16
Fecal fat levels | Baseline, Week 6, Week 12, Week 16
Fecal bile salt levels | Baseline, Week 6, Week 12, Week 16
Serum insulin/C-peptide | Baseline, Week 6, Week 12, Week 16

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Health Science and Technology, Aalborg University, Gistrup
  - Steno Diabetes Center Nordjylland, Gistrup

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive health information covered by the GDPR and cannot be made available outside the approved research team under Danish data protection regulations.

REFERENCES:
- [Background] Shen, X., Ma, C., Yang, Y., Liu, X., Wang, B., Wang, Y., Zhang, G., Bian, X., & Zhang, N. (2024). The Role and Mechanism of Probiotics Supplementation in Blood Glucose Regulation: A Review. https://doi.org/10.3390/foods13172719
- [Background] Kimura, I., Ozawa, K., Inoue, D., Imamura, T., Kimura, K., Maeda, T., Terasawa, K., Kashihara, D., Hirano, K., Tani, T., Takahashi, T., Miyauchi, S., Shioi, G., Inoue, H., & Tsujimoto, G. (2013). The gut microbiota suppresses insulin-mediated fat accumulation via the short-chain fatty acid receptor GPR43. Nature Communications, 4. https://doi.org/10.1038/NCOMMS2852,
- [Background] Dedrick, S., Sundaresh, B., Huang, Q., Brady, C., Yoo, T., Cronin, C., Rudnicki, C., Flood, M., Momeni, B., Ludvigsson, J., & Altindis, E. (2020). The Role of Gut Microbiota and Environmental Factors in Type 1 Diabetes Pathogenesis. Frontiers in Endocrinology, 11, 513621. https://doi.org/10.3389/FENDO.2020.00078/XML/NLM
- [Background] Abbasi, B., Mirlohi, M., Daniali, M., & Ghiasvand, R. (2018). Effects of probiotic soy milk on lipid panel in type 2 diabetic patients with nephropathy: A double-blind randomized clinical trial. Progress in Nutrition, 20(2-S), 70-78. https://doi.org/10.23751/PN.V20I2-S.5342
- [Background] Morshedi, M., Saghafi-Asl, M., & Hosseinifard, E. S. (2020). The potential therapeutic effects of the gut microbiome manipulation by synbiotic containing-Lactobacillus plantarum on neuropsychological performance of diabetic rats. Journal of Translational Medicine, 18(1). https://doi.org/10.1186/S12967-019-02169-Y,
- [Background] Keleszade, E., Kolida, S., & Costabile, A. (2022). The cholesterol lowering efficacy of Lactobacillus plantarum ECGC 13110402 in hypercholesterolemic adults: a double-blind, randomized, placebo controlled, pilot human intervention study. Journal of Functional Foods, 89, 104939. https://doi.org/10.1016/J.JFF.2022.104939
- [Background] Costabile, A., Buttarazzi, I., Kolida, S., Quercia, S., Baldini, J., Swann, J. R., Brigidi, P., & Gibson, G. R. (2017). An in vivo assessment of the cholesterol-lowering efficacy of Lactobacillus plantarum ECGC 13110402 in normal to mildly hypercholesterolaemic adults. https://doi.org/10.1371/journal.pone.0187964